CLINICAL TRIAL: NCT04573192
Title: A Study to Evaluate the Safety and Efficacy of the Tumor-targeting Human Antibody-cytokine Fusion Protein L19TNF Plus Lomustine in Patients With Glioblastoma at First Progression
Brief Title: A Study to Evaluate Safety and Efficacy of L19TNF Plus Lomustine in Patients With Glioblastoma at First Progression
Acronym: GLIOSTAR
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Philogen S.p.A. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PH-L19TNFCCNU-02/20
Record Dates: First submitted 2020-09-25; First posted 2020-10-05 (Actual); Last update posted 2024-04-08 (Actual); Status verified 2024-04

CONDITIONS: Glioblastoma
MeSH Terms: conditions — Glioblastoma | interventions — Lomustine

STUDY DESIGN:
Intervention Model Description: Open label phase I/II study in subjects with glioblastoma at first progression.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Phase 1 part: Dose Finding (Experimental): Phase I part:
  Dose Finding Patients will be treated in cohorts according to a traditional 3+3 design with lomustine on Day 1 and L19TNF on Days 1, 3 and 5, and on Days 22, 24 and 26, of a 42-days cycle at different dose levels.
  The RD will be confirmed following a traditional 3+3 design.
  Cohort 1: 10 µg /kg L19TNF i.v. plus 90 mg/m2 lomustine Cohort 2: 10 µg /kg L19TNF i.v. plus 110 mg/m2 lomustine Cohort 3: 13 µg /kg L19TNF i.v. plus 110 mg/m2 lomustine
  The dose of 13 ug/kg L19TNF will be declared the RD in case none of three or not more than one out of 6 patients experienced a DLT. Dose limiting toxicity will be assessed during the dose-escalation from Day 1 through Day 42 after the first administration of lomustine and study drug (Cycle 1). Not more than 2 patients might be treated simultaneously in Cycle 1.
  Interventions: Drug: L19TNF; Drug: Lomustine
- Phase II part: Signal Seeking (Experimental): 118 Patients will be randomized 1:1 and treated with either lomustine on day 1 and L19TNF on Days 1, 3 and 5, and on Days 22, 24, and 26 of a 42-days cycle at the RD established in the phase I part of the study or with lomustine on day 1 of a 42-days cycle.
  * Treatment Arm 1: L19TNF plus Lomustine
  * Treatment Arm 2: Lomustine
  Interventions: Drug: L19TNF; Drug: Lomustine

INTERVENTIONS:
Drug: L19TNF — Cohort 1: 10 µg /kg L19TNF i.v. plus 90 mg/m2 lomustine Cohort 2: 10 µg /kg L19TNF i.v. plus 110 mg/m2 lomustine Cohort 3: 13 µg /kg L19TNF i.v. plus 110 mg/m2 lomustine
  Other Names: onfekafusp alfa
Drug: Lomustine — Cohort 1: 10 µg /kg L19TNF i.v. plus 90 mg/m2 lomustine Cohort 2: 10 µg /kg L19TNF i.v. plus 110 mg/m2 lomustine Cohort 3: 13 µg /kg L19TNF i.v. plus 110 mg/m2 lomustine

SUMMARY:
Glioblastomas are the most common and most aggressive primary brain tumors in adults. The prognosis is poor despite multimodal therapy with surgery, radiotherapy and chemotherapy. Therefore, novel treatments are urgently needed.

L19TNF is a fully human fusion protein consisting of human tumor necrosis factor (TNF)-α fused to the L19 antibody in scFv format, specific to the extra-domain B of fibronectin. TNF not only induces apoptosis or necrosis in certain target cells, but also exerts inflammation and immunity. L19TNF selectively delivers TNF to the tumor site to spare normal tissues from undesired toxicity. Preclinical experiments with L19TNF have demonstrated tumor growth retardation in various mouse tumor models including models of glioma.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female, age ≥18.
2. Patients with histologically confirmed glioblastoma at unequivocal first recurrence or progression according to RANO criteria.
3. MGMT promotor methylation status known
4. IDH wildtype.
5. Patients may have undergone surgery for recurrence.
6. For operated patients: The histological report must document glioblastoma recurrence and a new MRI will need to be done at 3-5 weeks after surgery (directly before study treatment start). Study treatment will need to start minimum 4 weeks to maximum 6 weeks after surgery.
7. Karnofsky Performance Status (KPS) ≥ 70%.
8. Documented negative test for HIV-HBV-HCV. For HBV serology, the determination of HBsAg and anti-HBcAg Ab is required. In patients with serology documenting previous exposure to HBV, negative serum HBV-DNA is required. For HCV, HCV-RNA or HCV antibody test is required. Subjects with a positive test for HCV antibody but no detection of HCV-RNA indicating no current infection are eligible.
9. Female patients: female patients must be either documented not Women Of Childbearing Potential (WOCBP)* or must have a negative pregnancy test within 14 days of starting treatment. Additionally WOCBP must agree to use, from the screening to 6 months following the last study drug administration, highly effective contraception methods, as defined by the "Recommendations for contraception and pregnancy testing in clinical trials" issued by the Head of Medicine Agencies' Clinical Trial Facilitation Group (www.hma.eu/ctfg.html) and which include, for instance, progesterone-only or combined (estrogen- and progesterone-containing) hormonal contraception associated with inhibition of ovulation, intrauterine devices, intrauterine hormone-releasing systems, bilateral tubal occlusion or vasectomized partner.

   Male patients: male subjects able to father children must agree to use two acceptable methods of contraception throughout the study (e.g. condom with spermicidal gel). Double-barrier contraception is required.
10. Personally signed and dated informed consent document indicating that the subject has been informed of all pertinent aspects of the study.
11. Willingness and ability to comply with the scheduled visits, treatment plan, laboratory tests and other study procedures.

    * Women of childbearing potential are defined as females who have experienced menarche, are not postmenopausal (12 months with no menses without an alternative medical cause) and are not permanently sterilized (e.g., tubal occlusion, hysterectomy, bilateral oophorectomy, or bilateral salpingectomy).

Exclusion Criteria:

1. Prior treatment for glioblastoma at recurrence, except surgery.
2. Surgical resection or biopsy of glioma within 4 weeks of the start of study treatment.
3. Inability to undergo contrast-enhanced MRI.
4. Prior treatment with lomustine.
5. Known history of allergy to TNF or lomustine, any excipient in the study medication or any other intravenously administered human proteins/peptides/antibodies.
6. Absolute neutrophil count (ANC) < 1.5 x 10^9/L; platelets < 100 x 10^9/L or haemoglobin (Hb) < 9.0 g/dl.
7. Chronically impaired renal function as indicated by creatinine clearance < 60 mL/min or serum creatinine > 1.5 ULN.
8. Inadequate liver function (ALT, AST, ALP ≥ 2.5 x ULN or total bilirubin ≥ 2.0 x ULN).
9. INR > 1.5 ULN.
10. Any severe concomitant condition which makes it undesirable for the patient to participate in the study or which could jeopardize compliance with the protocol, in the opinion of the investigator.
11. Active or history of autoimmune disease that might deteriorate when receiving an immuno-stimulatory agent, in the judgement of the investigator.
12. History within the last year of cerebrovascular disease and/or acute or subacute coronary syndromes including myocardial infarction, unstable or severe stable angina pectoris.
13. Heart insufficiency (> Grade II, New York Heart Association (NYHA) criteria).
14. Clinically significant cardiac arrhythmias or requiring permanent medication.
15. LVEF <55% or any other abnormalities observed during baseline ECG and echocardiogram investigations that are considered as clinically significant by the investigator. Subjects with current or a history of QT/QTc prolongation are excluded.
16. Uncontrolled hypertension.
17. Known arterial aneurism at high risk of rupture.
18. Ischemic peripheral vascular disease (Grade IIb-IV according to Leriche-Fontaine classification).
19. Medically documented history of or active major depressive episode, bipolar disorder (I or II), obsessive-compulsive disorder, schizophrenia, a history of suicidal attempt or ideation, or homicidal ideation (e.g. risk of doing harm to self or others), or patients with active severe personality disorders.
20. Anxiety ≥ CTCAE Grade 3.
21. Severe diabetic retinopathy such as severe non-proliferative retinopathy and proliferative retinopathy.
22. Major trauma including major surgery (such as abdominal/cardiac/thoracic surgery) within 4 weeks of administration of study treatment.
23. Known history of tuberculosis.
24. Pregnancy or breast feeding.
25. Requirement of chronic administration of high dose corticosteroids or other immunosuppressant drugs. Subjects must have been either off corticosteroids, or on a stable or decreasing dose ≤ 4 mg daily dexamethasone (or equivalent) for 7 days prior to start of treatment. Limited or occasional use of corticosteroids to treat or prevent acute adverse reactions is not considered an exclusion criterion.
26. Presence of active and uncontrolled infections or other severe concurrent disease, which, in the opinion of the investigator, would place the patient at undue risk or interfere with the study.
27. Concurrent malignancies unless the patient has been disease-free without intervention for at least 2 years.
28. Growth factors or immunomodulatory agents within 7 days prior to the administration of study treatment.
29. Serious, non-healing wound, ulcer, or bone fracture.
30. Anticoagulation therapy with P2Y12 antagonists (e.g., clopidogrel, ticagrelor) and vitamin K antagonists (e.g., phenprocoumon, warfarin).
31. Requirement of concurrent use of other anti-cancer treatments or agents other than study medication.
32. Any live vaccination within 4 weeks prior to treatment or plan to receive live vaccination during the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 142 (Estimated)
Dates: Start 2021-02-19 (Actual); Primary Completion 2025-03 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
For Phase 1: DLT | For Cohort 1 to Cohort 3 from Day 1 to Day 42 after the first administration of lomustine and study drug (Cycle 1)
  Occurrence of dose limiting toxicity (DLT) assessed by frequency and grade of adverse events (AE) according to CTCAE v.5.0.
For Phase 2: Overall Survival | From beginning of treatment to 12 months
  Overall survival (OS) rate

SECONDARY OUTCOMES:
PFS | From the date of enrollment to the date of progression or death for any cause, whichever came first, assessed up to 52 weeks
  Progression-free survival (PFS) based on iRANO criteria and a standardized MRI protocol will be assessed for all enrolled subjects.
PFS-rate at 6 months | From the date of enrollment to the date of progression or death for any cause, whichever came first, assessed up to 6 months
  Progression-free survival (PFS) based on iRANO criteria and a standardized MRI protocol will be assessed for all enrolled subjects
OS-rate at 12 months | From beginning of treatment to 12 months
Adverse Events (AE) | Throughout study completion for each patient, a maximum of 52 weeks for each patient
  Safety of administration of L19TNF, through an assessed by Common Toxicity Criteria (version 5.0, CTCAE)
Serious Adverse Events (AE) | Throughout study completion for each patient, a maximum of 52 weeks for each patient
  Safety of administration of L19TNF, assessed by Common Toxicity Criteria (version 5.0, CTCAE)
Safety (DILI) | Throughout study completion for each patient, a maximum of 52 weeks for each patient
  Evaluation of possible Drug Induce Liver Injury, caused by L19TNF, assessed by Common Toxicity Criteria (version 5.0, CTCAE)

CONTACTS AND LOCATIONS:
Locations (15):
- France (3):
  - Hôpital Neurologique Pierre Wertheimer, Bron
  - Hôpital Saint Louis, Paris
  - Sorbonne University, AP-HP, Paris brain institute, Paris
- Germany (4):
  - University Hospital Bonn, Bonn
  - University Hospital Köln, Cologne
  - Klinikum rechts der Isar, München
  - Universitatsklinikum Tubingen, Tübingen
- Italy (5):
  - Azienda USL di Bologna IRCCS delle Scienze Neurologiche di Bologna, Bologna
  - Fondazione IRCCS Istituto Neurologico Carlo Besta, Milan
  - Istituto Oncologico Veneto IRCCS, Padua
  - Azienda Ospedaliero-Universitaria Senese Policlinico Le Scotte, Siena
  - AOU Città della Salute e della Scienza di Torino, Torino
- Switzerland (3):
  - Inselspital Universitätsklinik für Medizinische Onkologie Bern, Bern
  - Centre Hospitalier Universitaire Vaudois (CHUV), Lausanne
  - Universitatspital Zurich - Klinik fur Neurologie & Hirntumorzentrum, Zurich

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Look T, Puca E, Buhler M, Kirschenbaum D, De Luca R, Stucchi R, Ravazza D, Di Nitto C, Roth P, Katzenelenbogen Y, Weiner A, Rindlisbacher L, Becher B, Amit I, Weller M, Neri D, Hemmerle T, Weiss T. Targeted delivery of tumor necrosis factor in combination with CCNU induces a T cell-dependent regression of glioblastoma. Sci Transl Med. 2023 May 24;15(697):eadf2281. doi: 10.1126/scitranslmed.adf2281. Epub 2023 May 24. PMID 37224228